CLINICAL TRIAL: NCT03393338
Title: Diabetes Interprofessional Team to Enhance Adherence to Medical Care
Acronym: DM I-TEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: University of the Sciences in Philadelphia (Other)
Responsible Party: Principal Investigator, Barry Rovner, Professor, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4100077081
Record Dates: First submitted 2017-12-31; First posted 2018-01-08 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Diabetes
Keywords: Diabetes; African American; Emergency Department visits
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DM I-TEAM (Experimental): DM I-TEAM is a home-based behavioral intervention that involve 9 treatment visits with a community health worker (CHW) over 12 months. During the treatment visits, the CHW provides culturally-relevant diabetes education, and facilitates telehealth visits with a diabetes nurse educator and participants' primary care physicians (PCPs). In addition, a clinical pharmacist reviews participants' medication regimens to identify potentially inappropriate medications (PIMS), and to simply regimens when indicated to facilitate medication adherence.
  Interventions: Behavioral: DM I-TEAM
- Usual Medical Care (No Intervention): Usual medical care

INTERVENTIONS:
Behavioral: DM I-TEAM — DM I-TEAM is a home-based behavioral intervention that involve 9 treatment visits with a community health worker (CHW) over 12 months. During the treatment visits, the CHW provides culturally-relevant diabetes education, and facilitates telehealth visits with a diabetes nurse educator and participants' primary care physicians (PCPs). In addition, a clinical pharmacist reviews participants' medication regimens to identify potentially inappropriate medications (PIMS), and to simply regimens when indicated to facilitate medication adherence.
  Arms: DM I-TEAM

SUMMARY:
The overall goal of this randomized controlled trial is to test the efficacy of DM I-TEAM (Diabetes Interprofessional Team to Enhance Adherence to Medical Care) to reduce emergency department (ED) visits and hospitalizations over 12 months in older African Americans (AAs) with diabetes mellitus (DM). DM I-TEAM is a multidisciplinary behavioral intervention that comprises a community health worker (CHW), the participant's primary care physician (PCP), a diabetes nurse educator, and a clinical geriatric pharmacist. In DM I-TEAM, the CHW conducts in-home sessions to: (1) provide diabetes education, (2) facilitate adherence to diabetes self-management behaviors (e.g., medication adherence glucose monitoring, diet, exercise); and (3) build trust between patients and their primary care team. This is accomplished by: (1) using culturally relevant diabetes educational materials; (2) facilitating telehealth visits with the participant's PCP and the diabetes nurse educator via JeffConnect; and (3) having the study pharmacist review participants' medication regimens to identify potentially inappropriate medications, simplify medication regimens if possible, and to reduce medication side effects.

DETAILED DESCRIPTION:
AAs have twice the rate of DM as Whites, and worse glycemic control, less optimal medication regimens, and less trust in the medical system. These disparities contribute to why AAs with DM are more likely to go blind, lose limbs, require dialysis, develop dementia, and die than Whites. These disparities, in turn, reflect racial differences in education, income, health literacy, cultural beliefs, experiences of discrimination, and social adversity, which can lead to: 1) poor glycemic control; 2) suboptimal medication use; and 3) mistrust in medical care. DM I-TEAM addresses these 3 factors, which often precipitate ED and hospital care, using a culturally relevant, multidisciplinary team treatment approach to reduce the need for high acuity medical care, and equip underserved AAs with DM with the knowledge and skill to gain the benefits of high quality medical care that is otherwise available to everyone. Our approach applies currently available treatment elements in a culturally-relevant way to create a more equitable health landscape. Our immediate goal is to engage a high-risk population in treatment that can be trusted; that recognizes the realities of their lives (e.g., financial insecurity); that improves the quality of the medication they take, and that builds their self-efficacy to manage DM. The intermediate goal is to prevent untoward medical events that necessitate ED or hospital care. The long-term goal is to reverse the pernicious racial disparities that now characterize healthcare in the U.S. DM I-TEAM can achieve these goals by getting the right care to the right patient at the right time. DM I-TEAM is the right care because its leverages existing resources in a new way to improve health outcomes in AAs with DM. AAs with DM are the right patients because many have poorly controlled DM, take suboptimal medications, and face treatment barriers, often social in nature. Now is the right time, as the population becomes more racially diverse, healthcare costs increase, and demand for safety, quality, and value intensify. In these ways DM I-TEAM is right for American healthcare, bringing us closer to Healthy People 2020's twin goals of reducing the personal and societal costs of DM, and achieving health equity for all.

DM I-TEAM takes a dynamic team approach to diabetes management whereby the primary care physician, the study pharmacist, the diabetes educator, and the CHW collaborate to build patient trust, encourage diabetes self-management, and optimize medication regimens. Each member of the team plays a pivotal role in identifying important information that prevents effective diabetes management, and then works together to provide multi-layered support to patients. The roles of each team member are as follows:

CHW: The CHW extends clinic-based care into participants' homes to strengthen patient/provider relationships, customize diabetes education, and develop tailored treatment plans. The CHW facilitates telemedicine visits with the PCP and diabetes educator to build trust in the health care system by increasing participants' access to their care team. The quality and content of these visits is enhanced by CHW-provided information about the participant's life situation (e.g., family circumstances, barriers to optimal diabetes self-management, home environment), and current self-management practices and beliefs. There will be 6 90 minute in-home CHW sessions within 3 months of randomization (telemedicine sessions will occur during 3 of these visits). Booster sessions will occur 5, 7, and 11 months after randomization. During these visits, the CHW will (1) reinforce the diabetes treatment plan articulated by the PCP, (2) gather information regarding barriers to diabetes self-management behaviors and communicate them to the team; (3) inform the team of the participant's health-related questions/issues; (4) provide culturally-relevant diabetes education using appropriate educational materials; (5) work with the participant to formulate and execute diabetes Action Plans using the principles of Behavioral Activation (BA); and (6) communicate the participant's progress with their Action Plans to the team. BA is a behavioral technique based on reinforcement theory that is used to help people overcome avoidant tendencies through goal setting, activity scheduling, and graded task assignment. BA was originally developed to treat depression. Our research has demonstrated that BA can successfully facilitate diabetes self-management. The DM I-TEAM treatment manual (which is already developed but will be refined during the study start-up phase) describes each session in detail, and includes scripts and didactics for the CHW interventionist. The manual is not included in this grant submission due to space limitations. At each session, the CHW educates participants to contact the ED (either by phone or by patient portal) prior to presenting for services. Participants are given "emergency kits" that contain glucometers and related supplies and glucose tablets. The ED physician may recommend that participant's test their glucose and treat hypoglycemia prior to or instead of reporting to the ED.

PCP: The PCP provides diabetes care as per standard practice, but care is supplemented with input from the pharmacist and the CHW, and with telemedicine visits. The PCP optimizes medication regimens based on pharmacist recommendations. As the course of treatment progresses, the PCP reinforces Action Plans with the participant during clinic visits.

Pharmacist: With information gathered by the CHW and from the participant's electronic medical records (EMR), the pharmacist performs a comprehensive evaluation of the participant's medications to identify medications that are contraindicated in older patients, are not being taken as prescribed, are being taken incorrectly, are improperly dosed, or may be causing undesirable side effects. Based on her assessment, the pharmacist may recommend that the PCP modify the current medication regimen.

Diabetes Educator: The diabetes educator provides telemedicine visits to supplement diabetes education provided by the CHW, answer participants' questions, and reinforce medication adherence.

ELIGIBILITY:
Inclusion Criteria:

1. African American race
2. Age ≥ 35 years; When first proposed the age criterion was 60 or older; it was later modified to 35 and older
3. Type 1 or 2 DM
4. A DM-related cause for the ED visit (i.e., hyperglycemia/hypoglycemia, diabetic ketoacidosis, chest pain, skin or soft tissue infection, diabetic neuropathy, retinopathy, urinary tract infection/pyelonephritis/acute renal injury, requesting DM medication refill) OR an hemoglobin A1c of 7.0% or greater within the past 30 days

Exclusion Criteria:

1. Evidence of cognitive and functional decline suggestive of dementia.
2. Anti-dementia medication use
3. Life expectancy less than one year (in the opinion of the evaluating ED physician)
4. DSM-V psychiatric disorders other than anxiety or depression (as per EMR)
5. Intoxicated
6. Suicidal
7. In police custody or currently incarcerated
8. Undergoing medical clearance for a detox center or any involuntary court or magistrate order
9. Lives in assisted living, currently in a rehabilitation facility (other than Jefferson), lives in a nursing home or skilled nursing facility
10. Pregnant

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of emergency room visits and hospitalizations over 12 months | 12 months
  The primary efficacy analysis will consider the number of incident diabetes-related ED visits and/or hospitalizations (i.e., an "event") over 12 months after the index ED visit. Each ED visit or hospitalization is counted as a single event (although an ED visit that leads to a hospitalization is counted once). ED visits and hospitalization will be ascertained through chart reviews and subject self-report.

SECONDARY OUTCOMES:
hemoglobin A1c | 12 months
  Subjects will have their hemoglobin A1c tested using a point of care test.
Potentially Inappropriate Medications (PIMS) | 12 months
  PIMS will be assessed via chart review by a clinical pharmacist.
Physician Trust | 12 months
  Physician trust will be assessed with the Multidimensional Trust in Health Care Systems. This 17-item scale measures trust in physicians (e.g., "I trust my doctor's judgment"); health payers (e.g., "Healthcare payers are good at what they do"); and health care institutions (e.g., "Healthcare institutions provide high quality care").

CONTACTS AND LOCATIONS:
Overall Officials: Barry Rovner, MD, Principal Investigator — Thomas Jefferson Uinversity
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rovner BW, Casten R, Chang AM, Hollander JE, Leiby BE, Nightingale G, Pizzi L, Herres J, White N, Kelley M, Rising K. Interprofessional Intervention to Reduce Emergency Department Visits in Black Individuals with Diabetes. Popul Health Manag. 2023 Feb;26(1):46-52. doi: 10.1089/pop.2022.0216. Epub 2023 Feb 6. PMID 36745390
- [Derived] Rovner BW, Casten RJ, Chang AM, Hollander JE, Rising K. Mistrust, Neighborhood Deprivation, and Telehealth Use in African Americans with Diabetes. Popul Health Manag. 2021 Dec;24(6):699-700. doi: 10.1089/pop.2021.0094. Epub 2021 May 17. PMID 34000211
- [Derived] Rovner BW, Casten RJ. Medication Beliefs and Depression in African Americans With Diabetes. Am J Geriatr Psychiatry. 2021 Dec;29(12):1296-1297. doi: 10.1016/j.jagp.2021.03.011. Epub 2021 Apr 9. No abstract available. PMID 33994087
- [Derived] Rovner BW, Casten RJ. Emergency department visits in African Americans with mild cognitive impairment and diabetes. J Diabetes Complications. 2021 May;35(5):107905. doi: 10.1016/j.jdiacomp.2021.107905. Epub 2021 Mar 16. PMID 33752964
- [Derived] Rovner BW, Casten RJ. Discordant health beliefs and telehealth use in African Americans with diabetes. J Am Geriatr Soc. 2021 Jun;69(6):1684-1686. doi: 10.1111/jgs.17081. Epub 2021 Mar 5. No abstract available. PMID 33675034
- [Derived] Rovner BW, Casten RJ, Chang AM, Hollander JE, Kelley M, Rising KL. Cognitive Deficits in African Americans With Diabetes in an Emergency Department. Am J Geriatr Psychiatry. 2020 Apr;28(4):503-504. doi: 10.1016/j.jagp.2019.07.018. Epub 2019 Aug 6. No abstract available. PMID 31477457